CLINICAL TRIAL: NCT05526807
Title: Feasibility Studies to Investigate the Role of Ursodeoxycholic Acid in the Prevention of Recurrence of C. Difficile Infection
Brief Title: Ursodeoxycholic Acid in C. Difficile Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17GA025
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Clostridioides Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ursodeoxycholic acid (Experimental): Only one arm - subjects receiving ursodeoxycholic acid
  Interventions: Drug: Ursodeoxycholic acid

INTERVENTIONS:
Drug: Ursodeoxycholic acid — Oral

SUMMARY:
The primary objective of the study is to assess tolerability and adherence to treatment with ursodeoxycholic acid

ELIGIBILITY:
Inclusion Criteria:

* Completion of a course of antibiotic treatment for C. difficile infection within the previous 7 days

Exclusion Criteria:

* • Pregnant or Breast-feeding

  * Gall bladder inflammation
  * Frequent episodes of biliary colic
  * Occlusion of the common bile duct or cystic duct
  * Active small intestinal inflammation
  * Previous resection of distal small intestine
  * Treatment with bile salt binding agents, ciclosporin or ciprofloxacin
  * Diarrhoea (from any cause) at study initiation
  * hypersensitivity to bile acids or any excipient of the formulation
  * Life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
To assess tolerability to oral ursodeoxycholic acid | 6 weeks
  Assess for side effects

SECONDARY OUTCOMES:
To determine recurrence of C. difficile infection in those able to take ursodeoxycholic acid | 12 weeks
  Recurrence of C. difficile infection to be confirmed by stool test for toxin(s)

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom